CLINICAL TRIAL: NCT02666001
Title: A Phase 1, Open-Label, Drug-Drug Interaction Study Between Methadone and BMS-663068; and Between Buprenorphine/Naloxone and BMS-663068
Brief Title: A Study to Assess the Drug-drug Interaction of BMS 663068 With Methadone and Also With Buprenorphine/Naloxone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 206216; AI438-068 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2016-01-06; First posted 2016-01-28 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — fostemsavir; Methadone; Buprenorphine; norbuprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (BMS-663068+methadone) (Experimental): Effect of multiple doses of BMS-663068, 600mg ER on the exposure of methadone
  Interventions: Drug: BMS-663068; Drug: Methadone
- Part 2 (BMS-663068+buprenorphine and norbuprene) (Experimental): Effect of multiple doses of BMS-663068, 600mg ER on the exposure of buprenorphine and norbuprenorphine
  Interventions: Drug: BMS-663068; Drug: Buprenorphine and Norbuprenorphine

INTERVENTIONS:
Drug: BMS-663068 — BMS-663068
Drug: Methadone — Methadone
  Arms: Part 1 (BMS-663068+methadone)
Drug: Buprenorphine and Norbuprenorphine — Buprenorphine and Norbuprenorphine
  Arms: Part 2 (BMS-663068+buprenorphine and norbuprene)

SUMMARY:
The study is being conducted to assess the effect of multiple doses of BMS-663068 on the exposure of methadone in subjects on a stable dose of methadone, and the exposure of buprenorphine and norbuprenorphine in subjects on a stable dose of buprenorphine and norbuprenorphine.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Target population: Subjects on methadone maintenance therapy (for inclusion in Part 1) or buprenorphine and norbuprenorphine maintenance therapy (for inclusion in Part 2), who have been reliably participating in an oral methadone or buprenorphine and norbuprenorphine program and who are on a stable dose for at least 30 days prior to study screening
3. Male and Female Subjects with body mass index of 18 to 34 kg/m2, inclusive
4. Women of child bearing potential (WOCBP) with negative serum or urine pregnancy test and must not be breastfeeding
5. Men and WOCBP must agree to follow instructions for contraception

Exclusion Criteria:

1. History of any chronic or acute illness, gastrointestinal disease, smoking and alcohol abuse
2. Any Gastrointestinal (GI) surgery within 4 weeks of study drug administration that could affect its absorption
3. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations beyond what is consistent with the target population.
4. History of allergy to any drugs, BMS-663068, HIV attachment inhibitors, or related compounds

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2016-06-29 (Actual); Study Completion 2016-06-29 (Actual)

PRIMARY OUTCOMES:
Cmax for Methadone (Part 1) and buprenorphine and norbuprenorphine (Part 2) | Days 1 to 10
AUC(TAU) for Methadone (Part 1) and buprenorphine and norbuprenorphine (Part 2) | Days 1 to 10

SECONDARY OUTCOMES:
Incidence of Adverse events (AEs), serious AEs (SAEs), and AEs leading to discontinuation. | For AEs, Days 1 to 10; for SAEs, Screening, Days 1 to 10 and up to 30 days post discontinuation of dosing

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (2):
- United States (2):
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Overland Park, Kansas

IPD SHARING:
Plan to Share IPD: No